CLINICAL TRIAL: NCT02931175
Title: An Open-label, Multi-center, Randomized, Phase II Study of the Safety,Efficacy and Bioactivity of Two Dose Regimens of Subcutaneous Injections of ACTH Gel in Patients With Non-infectious Uveitis
Brief Title: ACTH as A Re-emerging theRapy for Uveitis (The ACTHAR Study)
Acronym: ACTHAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Quan Dong Nguyen (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor-Investigator, Quan Dong Nguyen, MD, MSc (USA), Ocular Imaging Research and Reading Center
Organization: Ocular Imaging Research and Reading Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTHAR-01
Record Dates: First submitted 2016-10-06; First posted 2016-10-12 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2018-09

CONDITIONS: Uveitis
Keywords: ACTH gel; Non-Infectious Uveitis; ACTHAR; Posterior Uveitis; Intermediate Uveitis; Pan Uveitis; Uveitis
MeSH Terms: conditions — Uveitis; Uveitis, Posterior; Uveitis, Intermediate | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Mandatory twice a week (Mondays and Thursdays) treatment with SC ACTH gel 80 U/day starting at BL until month 6. Starting at month 6, the treatment will be administered on as needed basis, based on the retreatment criteria.
  Interventions: Drug: ACTH gel
- Group 2 (Experimental): Mandatory thrice a week (Mondays, Wednesdays, and Fridays) treatment with SC ACTH gel 80 U/day starting at BL until month 6. Starting at month 6, the treatment will be administered on as needed basis, based on the retreatment criteria.
  Interventions: Drug: ACTH gel

INTERVENTIONS:
Drug: ACTH gel — Starting at month 6, retreatment will be offered to study subjects who have demonstrated any level of response during the first 6 months and who meet any of these Retreatment Criteria listed below. Patients receiving retreatment will receive the dose that was assigned to them at randomization.
  Other Names: Corticotropin

SUMMARY:
The study aims to evaluate the potential role of ACTH gel in the management of non-infectious uveitis.

DETAILED DESCRIPTION:
Uveitis is a term used to describe a group of inflammatory disorders involving the uveal tract (iris, ciliary body and choroid). It is amongst the most common causes in the list of preventable cause of blindness in the developed world.

H.P. Acthar Gel is a highly purified sterile preparation of the adrenocorticotropic hormone (ACTH) gelatin to provide a prolonged release after intramuscular or subcutaneous (SC) injection.

ACTH is part of a group of molecules called melanocortins (MC) (ACTH, α, β, γ-MSH) that are produced, in human bodies, by breakdown of a common larger precursor called proopiomelanocortin (POMC). A very well-known anti-inflammatory mechanism of action of ACTH is the production glucocorticoids by stimulating the adrenal glands. ACTH has also been shown to bind with all five melanocortin receptors (MCRs). MCRs have a variety of roles including cortisol production and regulation of immune modulation by ACTH.

ACTHAR is an open-label, multi-center, randomized, phase II study to evaluate the effect of two dose regimens of repeated SC injections of ACTH gel in patients with active non-infectious intermediate, posterior, or pan-uveitis followed over a period of 12 months.

ACTHAR study will be conducted at up to 7 clinical sites in USA. The study will be coordinated by the Ocular Imaging Research and Reading Center (OIRRC), which will serve as the coordinating and reading center for the ACTHAR Study.

The primary endpoint of the study will be at month 6, with an active, as-needed treatment extension phase from month 6 to month 12.

Thirty-six (36) patients with non-infectious intermediate, posterior, or pan-uveitis will be enrolled and randomized (1:1) to one of the two treatment arms:

1. Mandatory twice a week (Mondays and Thursdays) treatment with SC ACTH gel 80 U/day starting at BL until month 6. Starting at month 6, the treatment will be administered on as needed basis, based on the retreatment criteria.
2. Mandatory thrice a week (Mondays, Wednesdays, and Fridays) treatment with SC ACTH gel 80 U/day starting at BL until month 6. Starting at month 6, the treatment will be administered on as needed basis, based on the retreatment criteria.

Starting at month 6, retreatment will be offered to study subjects who have demonstrated any level of response during the first 6 months and who meet any of these Retreatment Criteria listed below. Patients receiving retreatment will receive the dose that was assigned to them at randomization.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for the study, patients will be required to meet the criteria of 1 of the 3 following disease cohorts:

1. Active disease and are receiving no treatment. Active disease is defined as having at least 1+ Vitreous Haze using the Standardized Uveitis Nomenclature (SUN) Working Group scale and/or at least 1+ Vitreous Cell Count using Foster & Vitale scale.
2. Active disease and are receiving prednisone ≥10 mg/day (or equivalent dose of another corticosteroid) or at least 1 other systemic immunosuppressant (all systemic immunosuppressants other than corticosteroids will be discontinued 30 days prior to the first administration of the study drug on Day 0). Patients receiving combination of prednisone ≥10 mg/day and at least one other systemic immunosuppressant are also eligible in this category.
3. Have inactive disease, defined as having <= 0.5+ Vitreous Haze OR <= 0.5+ Vitreous Cell Count (SUN scale), and are receiving prednisone ≥10 mg/day (or equivalent dose of another corticosteroid) or at least 1 other systemic immunosuppressant (all systemic immunosuppressants other than corticosteroids will be discontinued 30 days prior to the first administration of the study drug on Day 0). Patients receiving combination of prednisone ≥10 mg/day and at least one other systemic immunosuppressant are also eligible in this category.

Exclusion Criteria:

Subjects who have any of the following at the screening visit are not eligible for enrolment in this study:

1. Any significant ocular disease that could compromise vision in the study eye. These include, but are not limited to:

   * Diabetic retinopathy: proliferative diabetic retinopathy (PDR) or non-proliferative diabetic retinopathy (NPDR) that compromise the vision.
   * Age-related macular degeneration;
   * Myopic degeneration with active subfoveal choroidal neovascularization.
   * Advanced glaucoma status post trabeculectomy or tube/valve placement
2. Any of the following treatments within 90 days prior to Day 0 or anticipated use of any of the following treatments to the study eye:

   * Intravitreal injections (including but not limited to steroids or anti-vascular endothelial growth factors);
   * Posterior subtenon's steroids.
3. Intraocular surgery within 90 days prior to Day 0 in the study eye;
4. Capsulotomy within 30 days prior to Day 0 in the study eye;
5. Any known ocular surgery (including cataract extraction or capsulotomy) of the study eye anticipated within the first 180 days following Day 0;
6. Intraocular pressure(IOP) ≥25 mmHg in the study eye (glaucoma patients maintained on no more than 2 topical medications with IOP <25 mmHg are allowed to participate);
7. Pupillary dilation inadequate for quality stereoscopic fundus photography in the study eye;
8. Media opacity that would limit clinical visualization;
9. Presence of any form of ocular malignancy in the study eye, including choroidal melanoma;
10. History of herpetic infection in the study eye or adnexa;
11. Presence of known active or inactive toxoplasmosis in either eye;
12. Presence of ocular or periocular infection in either eye;
13. Participation in other investigational drug or device clinical trials within 30 days prior to Day 0, or planning to participate in other investigational drug or device clinical trials within 180 days following Day 0. This includes both ocular and non-ocular clinical trials.
14. Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following randomization.
15. Prior treatment with any cell-depleting therapies, including investigational agents or approved therapies, some examples are anti-cluster of differentiation (CD) 4, anti- cluster of differentiation (CD)5, anti-cluster of differentiation (CD) 3, anti-cluster of differentiation (CD)19 and anti-cluster of differentiation (CD)20.
16. Treatment with intravenous gamma globulin, plasmapheresis or Prosorba column within 6 months of baseline.
17. Immunization with a live/attenuated vaccine within 4 weeks prior to baseline.
18. Previous treatment with ACTHAR within 3 months of day 0 of study visit.
19. Any previous treatment with alkylating agents such as chlorambucil, or with total lymphoid irradiation.

    Exclusions for General Safety:
20. History of severe allergic or anaphylactic reactions to proteins of porcine origin.
21. Evidence of serious uncontrolled concomitant cardiovascular (including history of congestive heart failure, uncontrolled hypertension), nervous system (include myasthenia gravis), pulmonary (including obstructive pulmonary disease), renal, hepatic, endocrine (include uncontrolled diabetes mellitus, hypothyroidism), gastrointestinal disease (including history of or presence peptic ulcer disease, complicated diverticulitis, ulcerative colitis, or Crohn"s disease), Scleroderma or Osteoporosis.
22. Current liver disease as determined by principal investigator unless related to primary disease under investigation.
23. Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections (including but not limited to tuberculosis and atypical mycobacterial disease, Hepatitis B and C, and herpes zoster, but excluding fungal infections of nail beds).
24. Any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening.
25. Active Tuberculosis (TB) requiring treatment within the previous 3 years. Patients should be evaluated for latent and/or active TB within one month of the screening as part of the evaluation by the investigator to rule out infectious uveitis before referring the patient to the study. If positive, patients should be managed following local practice guidelines prior to initiating H.P. ACTHAR gel. Patients treated for TB with no recurrence in 3 years are permitted.
26. Primary or secondary immunodeficiency (history of or currently active)
27. Evidence of active malignant disease, malignancies diagnosed within the previous 5 years (including hematological malignancies and solid tumors, except basal and squamous cell carcinoma of the skin or carcinoma in-situ of the cervix uteri that has been excised and cured)
28. Pregnant women or nursing (breast feeding) mothers.
29. Patients with reproductive potential not willing to use an effective method of contraception.
30. History of alcohol, drug or chemical abuse within 1 year prior to screening.
31. Neuropathies or other conditions that might interfere with pain evaluation unless related to primary disease under investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Incidence of ocular adverse events (AEs) | Month 6
  The incidence and severity of ocular adverse events, as identified by eye examination.
Incidence of systemic adverse events (AEs) | Month 6
  The incidence and severity of systemic adverse events.

SECONDARY OUTCOMES:
Mean change from Baseline (BL) in vitreous haze (VH) | Month 6
  Mean change from BL in vitreous haze using the Standardization of Uveitis Nomenclature (SUN) scale.
Proportion of patients achieving a ≥ 1 and ≥ 2 step improvement or resolution of VH | Month 3, 6, 12
  The proportion of patients achieving a ≥ 1 and ≥ 2 step improvement or resolution of VH on SUN scale after therapy or at time of rescue.
Mean change from BL in graded anterior chamber cells | Month 3, 6, 12
  Mean change from BL in graded anterior chamber cells after therapy or at time of rescue.
Mean change from BL in Best Corrected Visual Acuity (BCVA) | Month 3, 6, 12
  Mean change from BL in BCVA using the ETDRS
Mean change in degree of inflammation | Month 3, 6, 12
  Mean change in degree of intermediate uveitis, retinal vasculitis, chorioretinitis, or other types of inflammation as documented at baseline compared to evaluation at month 6 and 12 after therapy or at time of rescue.
Mean change in leakage of disc. | Month 3,6, 12
  Mean change in leakage of disc
Change from Baseline in macular thickness | Month 3, 6, 12
  Change from Baseline in macular thickness as measured by Spectral Domain Optical Coherence Tomography (SD-OCT).
The proportion of patients who achieve a complete response in the study eye and discontinue prednisone. | Month 3, 6, 12
  The proportion of patients who achieve a complete response in the study eye and discontinue prednisone.
The proportion of patients who achieve a partial response in the study eye and discontinue prednisone. | Month 3, 6, 12
  The proportion of patients who achieve a partial response in the study eye and discontinue prednisone.
Proportion of patients achieving a ≥ 1 and ≥ 2 step improvement or resolution of VH | Month 12
  The proportion of patients achieving a ≥ 1 and ≥ 2 step improvement or resolution of VH on SUN scale after therapy or at time of rescue.
Mean change from BL in graded vitreous cells | Month 3, 6, 12
  Mean change from BL in graded vitreous cells after therapy or at time of rescue.
Mean change from BL in aqueous flare | Month 3, 6 12
  Mean change from BL in aqueous flare as measured by aqueous flare meter.
Mean change in leakage of vasculature | Month 3,6, 12
  Mean change in leakage of vasculature
Mean change in leakage of chorioretinal lesions | Month 3, 6, 12
  Mean change in leakage of chorioretinal lesions
Mean change in Leakage in Macula | Month 3, 6, 12
  Mean change in Leakage in Macula
Changes in OCTA | Months 3, 6, 12
  Changes in OCTA at various time points

CONTACTS AND LOCATIONS:
Overall Officials: Quan D Nguyen, MD MSc, Principal Investigator — Ocular Imaging Research and Reading Center
Locations (7):
- United States (7):
  - Retina Vitreous Associates, Medical Group, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Metropolitan Eye Research and surgery Institute, Waltham, Massachusetts
  - Retina Centers Professional Corporation - RCPC, Cleveland, Ohio
  - Retina Consultants of Houston, Bellaire, Texas
  - Texas Retina Assiciates, Dallas, Texas
  - TExas Retina Associates, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sadiq MA, Agarwal A, Hassan M, Afridi R, Sarwar S, Soliman MK, Do DV, Nguyen QD. Therapies in Development for Non-Infectious Uveitis. Curr Mol Med. 2015;15(6):565-77. doi: 10.2174/1566524015666150731103847. PMID 26238367
- [Background] Montero-Melendez T. ACTH: The forgotten therapy. Semin Immunol. 2015 May;27(3):216-26. doi: 10.1016/j.smim.2015.02.003. Epub 2015 Feb 26. PMID 25726511
- [Background] Durrani OM, Meads CA, Murray PI. Uveitis: a potentially blinding disease. Ophthalmologica. 2004 Jul-Aug;218(4):223-36. doi: 10.1159/000078612. PMID 15258410
- [Background] Lee K, Bajwa A, Freitas-Neto CA, Metzinger JL, Wentworth BA, Foster CS. A comprehensive review and update on the non-biologic treatment of adult noninfectious uveitis: part I. Expert Opin Pharmacother. 2014 Oct;15(15):2141-54. doi: 10.1517/14656566.2014.948417. PMID 25226529